CLINICAL TRIAL: NCT01294267
Title: PERcutaneous heModynamic Support With Impella 2.5 During Scar-related Ventricular Tachycardia Ablation
Acronym: PERMIT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, DIRECTOR CARDIAC ARRHYTHMIA SERVICE, PROFESSOR OF MEDICINE, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 10-1423; BRANY IRB-10-02-154-05 (Other: BRANY - Biomedical Research Alliance of New York, an institutional review board fully accredited by AAHRPP)
Record Dates: First submitted 2011-01-25; First posted 2011-02-11 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Radio Frequency Ablation; Percutaneous Left Ventricular Assist Device; Hemodynamic Management; Interventional Cardiac Procedure; Mechanical Cardiac Assistance; Intra-Aortic Balloon Pump; Coronary Intervention; Impella 2.5; Circulation Support system
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Circulatory Support System (Other): Percutaneous use of left ventricular assist device, Impella 2.5 Circulatory Support System to facilitate mapping and ablation of ongoing VT by maintaining near-normal hemodynamics, reducing myocardial workload and preservice organ perfusion.
  Interventions: Device: Circulatory Support System

INTERVENTIONS:
Device: Circulatory Support System — Femoral angiography will be performed, and if the anatomy is suitable, the femoral artery preclosure technique will be employed. The Impella 2.5 will be inserted through th femoral artery into the left ventricle. Anti-coagulation will be titrated to achieve a therapeutic ACT level. Organ perfusion and Hemodynamic data will be collected during simulated VTs and throughout the course of the case. The performance level of the device may be adjusted during the case to quantify hemodynamic effects
  Other Names: Impella 2.5 Circulatory Support system insertion

SUMMARY:
The purpose of this research study is to evaluate the safety and feasibility of the Impella 2.5 Circulatory Support System for use during mapping and ablation of ventricular tachycardia in the setting of Ventricular dysfunction.

DETAILED DESCRIPTION:
The Impella 2.5 is a percutaneous heart pump that will be used to provide partial circulatory support -. The Impella 2.5 is approved by the US Food and Drug Administration and is being tested to see if it helps keep the patient's blood pressure stable during the cardiac ablation procedure. The Impella 2.5 Circulatory Support System works by placing a small pump into the left pumping chamber of the heart which will then help the heart circulate blood throughout the body. The Impella 2.5 Circulatory Support system will be removed once the heart no longer needs help with the pumping action which can be at any time from just after the completion of the heart procedure up to several days post procedure as determined by physician.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 18 to 90 years
* catheter ablation of ventricular tachycardia
* Left Ventricular ejection fraction less than or equal to 40% or hypertrophic cardiomyopathy

Exclusion Criteria:

* Any reversible cause of VT [electrolyte derangements, medication related itc]
* Evidence of active, ongoing cardiac ischemia as the cause of VT
* Patients who have experienced any cerebral ischemic event including any TIA in the preceding one month
* Mural thrombus in left Ventricle
* Presence of mechanical aortic valve
* Severe Aortic Stenosis [orifice area of 2.0 cm2 or less] or moderate to severe aortic insufficiency
* Severe abnormalities of the aorta that would preclude Impella insertion, including aneurysms and extreme tortuosity or calcifications
* Liver dysfunction or markedly abnormal coagulation parameters [as defined by platelet count less than or equal to 50,000/ul]
* Any condition resulting in contraindication to anticoagulation [eg GI bleeding]
* Women who are known to be pregnant or have had a positive B-HCG test 7 days prior to procedure
* Patients whose life expectancy is less than one year
* Mental Impairment precluding patient or family from providing informed consent or completing the appropriate follow up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller MA, Dukkipati SR, Chinitz JS, Koruth JS, Mittnacht AJ, Napolitano C, d'Avila A, Reddy VY. Percutaneous hemodynamic support with Impella 2.5 during scar-related ventricular tachycardia ablation (PERMIT 1). Circ Arrhythm Electrophysiol. 2013 Feb;6(1):151-9. doi: 10.1161/CIRCEP.112.975888. Epub 2012 Dec 19. PMID 23255277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty consecutive patients with scar VT underwent ablation between Sept 2010 and July 2011.
Period: Overall Study
Arm/Group | Circulatory Support System
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Circulatory Support System
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 13
  More than one race | 0
  Unknown or Not Reported | 3
Hypertension [Count of Participants; unit: Participants] | 14
Chronic Kidney Disease [Count of Participants; unit: Participants] | 6
Diabetes Mellitus [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural Success
Description: Satisfactory hemodynamic status during the ablation procedure [during VT Mapping and Ablation Procedure], utilizing the Hemodynamic Support of Impella 2.5 Circulatory Support System
Time Frame: Inpatient Admission
Measure: Count of Participants; unit: Participants
Arm/Group | Circulatory Support System
Number analyzed (Participants) | 20
Participants
  Complete procedural sucess | 8
  Partial procedural sucess | 6

2. Secondary Outcome: Clinical Outcomes
Description: Morbidity and Mortality, as determined by clinical metrics and validated by tests during and immediately post VT Mapping and ablation procedure with cardiac monitoring in hospital and one Month [30 days] follow up telephone interview to assess symptoms, side effects and medication use.
Time Frame: 1 Month post ablation Follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Circulatory Support System
Number analyzed (Participants) | 20
Participants
  Death from any cause | 2
  Hospitalization for any cause | 5
  Sustained VT/ICD therapy | 4

3. Other Pre Specified Outcome: Safety Outcomes
Description: Acute Kidney Injury Network stage 1 kidney injury (ie, an absolute increase in serum creatinine of ≥0.3 mg/dL or percentage increase of 150%-200% from baseline.
  A decline in neurocognitive function, as defined by a decrease in MMSE ≥2 points from the baseline score, after the procedure.
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | Circulatory Support System
Number analyzed (Participants) | 20
Participants
  Acute kidney injury stage 1 | 3
  Postop cognitive dysfunction | 1

ADVERSE EVENTS:
Arm/Group | Circulatory Support System
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circulatory Support System (N=20)
Death (Cardiac disorders) | 2 (2) — death from any cause
Hospitalization (General disorders) | 5 (5) — hospitalization for any cause, within 30 days
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circulatory Support System (N=20)
Acute Kidney Injury (Renal and urinary disorders) | 3 (20) — an absolute increase in serum creatinine of ≥0.3 mg/dL or percentage increase of 150%-200% from baseline), and all resolved within 72 hours

LIMITATIONS AND CAVEATS:
The lack of a control group precludes drawing definitive conclusions between the lack of either statistically or clinically significant changes in perioperative markers of end-organ perfusion/function and the use of a pLVAD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes